CLINICAL TRIAL: NCT01578746
Title: Comparison Between Minimally Invasive Anterior Approach and Direct Lateral Approach in Total Hip Arthroplasty - A Prospective Randomized Trial
Brief Title: Comparison Between Anterior and Direct Lateral Approach in Total Hip Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 811398; 2011/2581 D (Other: Regioal Ethics Commitee Norway)
Record Dates: First submitted 2012-03-13; First posted 2012-04-17 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Coxarthrosis
Keywords: Coxarthrosis; Hip arthroplasty; Anterior approach; Direct lateral approach; Hardinge approach; Smith-Petersen approach; Osteoarthrosis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Direct lateral approach (Active Comparator): Patient operated using direct lateral approach.
  Interventions: Procedure: Direct lateral approach in total hip arthroplasty
- Anterior approach (Active Comparator): Patient operated using anterior approach.
  Interventions: Procedure: Anterior approach

INTERVENTIONS:
Procedure: Direct lateral approach in total hip arthroplasty — The use of direct lateral approach in total hip arthroplasty
  Other Names: Hardinge approach
  Arms: Direct lateral approach
Procedure: Anterior approach — The use of anterior approach in total hip arthroplasty
  Other Names: Smith-Petersen approach
  Arms: Anterior approach

SUMMARY:
In total hip arthroplasty several approaches can be used. The newly introduced minimally invasive anterior approach is supposed to cause less damage to tendons and muscles. At the same time there are reports that there are more complications when this approach is used. The direct lateral approach is the most used in Norway and is well documented. There are however those who postulate that there is to high risk of damage to the gluteus medius causing Trendelenburg gait. In the investigators hospital both the anterior and direct lateral approach is used with good result. The investigators main study hypothesis is that there is no difference between the use of anterior or direct lateral approach i total hip arthroplasty in regards to postoperative function and pain, complications, radiological finds (X-ray and MRI), markers for muscle damage (i.e CK-total) or other clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of coxarthrosis

Exclusion Criteria:

* Previous surgery on affected hip
* No mental disability preventing follow-up

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in function | 2 years
  Function of the operated hip will be evaluated after 3, 6, 12 and 24 months using Oxford Hip Score, Harris Hip Score and 6-minute-walk-test. Improvement in general health will be evaluated by using Eq-5D.

SECONDARY OUTCOMES:
Muscle damage | Day of operation and next four consecutive days
  CK-total is measured direct postoperativly and for the next four consequtive days. CRP is measured the first four postoperative days.
Pain | First four postoperative days
  Pain using Visual Analog Scale and the use of analgetics (converted to opioid equivalent doses) are recorded.
X-ray assessment | 3 and 12 months
  Placement of the acetabular component (inclination and version) and femoral stem (varus/valgus) and migration.
MRI | 3 and 12 months
  A subselection of about 40 patients will undergo MRI-scans preoperatively and after 3 and 12 months to assess tendon- and muscledamage.

CONTACTS AND LOCATIONS:
Overall Officials: Svein Andreas Svenningsen, M.D, Ph.D, Principal Investigator — Sorlandet Hospital HF
Locations (1):
- Sorlandet Hospital HF, Arendal, Norway